CLINICAL TRIAL: NCT02030821
Title: TXA (Tranexamic Acid) vs. Amicar (Aminocaproic Acid) in Total Knee and Hip Arthroplasty- Effectiveness, Safety, and Cost Analysis
Brief Title: TXA vs. Amicar in Total Knee and Hip Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00050108
Record Dates: First submitted 2014-01-06; First posted 2014-01-09 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Blood Loss; Hip Arthritis; Knee Arthritis
MeSH Terms: conditions — Hemorrhage | interventions — Aminocaproic Acid; Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (TXA) (Active Comparator): TXA will be administered as a 1 gm dose IV prior to the procedure then as a repeat dose of 1 gram at the time of wound closure. These doses are currently used at Duke for Total Knee Arthroplasties (TKAs) and Total Hip Arthroplasties (THAs) per standard of care by the orthopaedic team.
  All data needed for this study including blood loss, need for transfusion, preoperative and lowest postoperative hematocrit and hemoglobin, and complications will be collected during the hospitalization.
  Interventions: Drug: TXA
- Epsilon-aminocaproic acid (Amicar) (Active Comparator): Administered 5g in 250mL of IV normal saline over 15 minutes prior to the procedure and then an infusion of 5g at the time of wound closure. These doses are currently used at Duke for Total Knee Arthroplasties (TKAs) and Total Hip Arthroplasties (THAs) per standard of care by the orthopaedic team.
  All data needed for this study including blood loss, need for transfusion, preoperative and lowest postoperative hematocrit and hemoglobin, and complications will be collected during the hospitalization.
  Interventions: Drug: Amicar

INTERVENTIONS:
Drug: Amicar — Subjects randomized to receive Amicar will receive this during surgical intervention
  Other Names: Aminocaproic Acid
  Arms: Epsilon-aminocaproic acid (Amicar)
Drug: TXA — Subjects randomized to receive TXA will receive this during surgical intervention
  Other Names: Tranexamic Acid
  Arms: Tranexamic Acid (TXA)

SUMMARY:
The purpose of this study is to determine the relative effectiveness of two drug agents, Tranexamic acid (TXA) and aminocaproic acid (Amicar), that act through a similar mechanism of action. These agents are used to decrease blood loss that is a result of major surgery, like total joint arthroplasty. A secondary goal will be investigate the cost-analysis of total hospitalization. Both TXA and Amicar are both currently used in the care of patients undergoing total joint arthroplasty.

Subjects will be randomly assigned to the TXA or Amicar arm. All data needed for this study including blood loss, need for transfusion, preoperative and lowest postoperative hematocrit and hemoglobin, and complications will be collected during the hospitalization stay.

Our Hypothesis is that TXA and Amicar will have similar effectiveness in preventing intraoperative blood loss and the need for transfusion post-op than Amicar.

A detailed cost analysis will show that the overall cost of performing the operative procedure, including transfusions, OR time, and total costs associated with admission cost will be more decreased with Amicar as compared to TXA.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing to undergo primary total hip or knee arthroplasty

Exclusion Criteria:

* History of stents
* Myocardial infarction,
* Cerebrovascular accident or stroke
* Deep venous thrombus
* Pulmonary embolus
* Late onset color blindness
* Hypercoagulable state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2015-01; Primary Completion 2017-11-12 (Actual); Study Completion 2017-11-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consenting completed at PI and co-investigators' private offices, clinic and in preoperative center. Study staff approved by the IRB consent the patients. First patient enrolled in January 2015. Last patient enrolled on 11/12/17.
Pre-assignment Details: Patients were excluded from the trial after enrollment if their surgery was cancelled.
Groups:
- Tranexamic Acid (TXA) - Total Hip Arthroplasty; Tranexamic Acid (TXA) - Total Knee Arthroplasty: TXA will be administered as a 1 gm dose IV prior to the procedure then as a repeat dose of 1 gram at the time of wound closure. These doses are currently used at Duke for TKAs and THAs per standard of care by the orthopaedic team.
  All data needed for this study including blood loss, need for transfusion, preoperative and lowest postoperative hematocrit and hemoglobin, and complications will be collected during the hospitalization.
  TXA: Subjects randomized to receive TXA will receive this during surgical intervention
- Epsilon-aminocaproic Acid (Amicar) - Total Hip Arthroplasty; Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty: Administered 5g in 250mL of IV normal saline over 15 minutes prior to the procedure and then an infusion of 5g at the time of wound closure. These doses are currently used at Duke for TKAs and THAs per standard of care by the orthopaedic team.
  All data needed for this study including blood loss, need for transfusion, preoperative and lowest postoperative hematocrit and hemoglobin, and complications will be collected during the hospitalization.
  Amicar: Subjects randomized to receive Amicar will receive this during surgical intervention
Period: Overall Study
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Hip Arthroplasty | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty
Started | 48 | 46 | 78 | 74
Completed | 46 | 44 | 73 | 72
Not Completed | 2 | 2 | 5 | 2
Not completed — Physician Decision | 2 | 2 | 5 | 2

BASELINE CHARACTERISTICS:
Population: All subjects who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Hip Arthroplasty | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty | Total
Number analyzed (Participants) | 46 | 44 | 73 | 72 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 26 | 29 | 37 | 35 | 127
  >=65 years | 20 | 15 | 36 | 37 | 108
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 50 | 42 | 140
  Male | 19 | 23 | 23 | 30 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 45 | 44 | 72 | 72 | 233
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 15 | 18 | 46
  White | 38 | 36 | 57 | 52 | 183
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 2 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 44 | 73 | 72 | 235

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss Over Course of Stay (Intraoperative and Postoperatively Until Discharge)
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Measure: Median (Inter-Quartile Range); unit: milliliters
Groups:
- Epsilon-aminocaproic Acid (Amicar); Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty: Administered 5g in 250mL of IV normal saline over 15 minutes prior to the procedure and then an infusion of 5g at the time of wound closure. These doses are currently used at Duke for TKAs and THAs per standard of care by the orthopaedic team.
  All data needed for this study including blood loss, need for transfusion, preoperative and lowest postoperative hematocrit and hemoglobin, and complications will be collected during the hospitalization.
  Amicar: Subjects randomized to receive Amicar will receive this during surgical intervention
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty
Number analyzed (Participants) | 46 | 44 | 73 | 72
milliliters | 934.1 [722.6 to 1173.1] | 948.7 [755.6 to 1314.8] | 660.6 [514.4 to 979.7] | 891.2 [612.1 to 1202.7]
Statistical Analysis 1: Comparison: Tranexamic Acid (TXA) - Total Hip Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) vs Tranexamic Acid (TXA) - Total Knee Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty; Test type: Other; p < 0.05, Kruskal-Wallis

2. Primary Outcome: Number of Transfusions
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Measure: Number; unit: transfusions
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty
Number analyzed (Participants) | 46 | 44 | 73 | 72
transfusions | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Tranexamic Acid (TXA) - Total Hip Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) vs Tranexamic Acid (TXA) - Total Knee Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty; Test type: Other; p < 0.05, Chi-squared

3. Primary Outcome: Difference in Preoperative and Lowest Postoperative Hemoglobin
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Measure: Median (Inter-Quartile Range); unit: grams per deciliter
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty
Number analyzed (Participants) | 46 | 44 | 73 | 72
grams per deciliter | 2.4 [1.5 to 3.2] | 2.6 [2.0 to 3.0] | 1.9 [1.2 to 2.4] | 2.1 [1.6 to 2.8]
Statistical Analysis 1: Comparison: Tranexamic Acid (TXA) - Total Hip Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) vs Tranexamic Acid (TXA) - Total Knee Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty; Test type: Other; p < 0.05, Kruskal-Wallis

4. Secondary Outcome: Length of Hospitalization Stay
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty
Number analyzed (Participants) | 46 | 44 | 73 | 72
days | 2.5 [2 to 3] | 3 [2 to 3] | 3 [2 to 3] | 3 [2 to 3]
Statistical Analysis 1: Comparison: Tranexamic Acid (TXA) - Total Hip Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) vs Tranexamic Acid (TXA) - Total Knee Arthroplasty vs Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty; Test type: Other; p < 0.05, Kruskal-Wallis

5. Secondary Outcome: Cost of Hospitalization
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 5 days
Population: Data not collected.
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Within 90 days of surgery
Arm/Group | Tranexamic Acid (TXA) - Total Hip Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Hip Arthroplasty | Tranexamic Acid (TXA) - Total Knee Arthroplasty | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44 | 0/73 | 0/72
Serious Adverse Events (participants affected / at risk) | 3/46 | 0/44 | 3/73 | 0/72
Other Adverse Events (participants affected / at risk) | 3/46 | 1/44 | 1/73 | 1/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (TXA) - Total Hip Arthroplasty (N=46) | Epsilon-aminocaproic Acid (Amicar) - Total Hip Arthroplasty (N=44) | Tranexamic Acid (TXA) - Total Knee Arthroplasty (N=73) | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty (N=72)
Acute Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
NSTEMI (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Deep Infection (Infections and infestations) | 3 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tranexamic Acid (TXA) - Total Hip Arthroplasty (N=46) | Epsilon-aminocaproic Acid (Amicar) - Total Hip Arthroplasty (N=44) | Tranexamic Acid (TXA) - Total Knee Arthroplasty (N=73) | Epsilon-aminocaproic Acid (Amicar) - Total Knee Arthroplasty (N=72)
Superficial Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Hematoma/Seroma (General disorders) | 1 | 1 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT02030821/Prot_SAP_000.pdf